CLINICAL TRIAL: NCT04742244
Title: Evaluation of the Efficacy of Supplementation With Lemon Verbena Extract in Improving
Brief Title: Lemon Verbena Extract Oxidative Stress and Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chi-Chang Huang, PI, National Taiwan Sport University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00002
Record Dates: First submitted 2021-01-25; First posted 2021-02-08 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Muscle Injury; Muscle Soreness
Keywords: DOMS,; Lemon verbena
MeSH Terms: conditions — Myalgia | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 0 mg LVE/capsule, 2capsule/day, 14days
  Interventions: Dietary Supplement: maltodextrin
- Lemon Verbena extract (Experimental): 200 mg LVE/capsule, 2capsule/day, 14days
  Interventions: Dietary Supplement: Lvemon verbena extract

INTERVENTIONS:
Dietary Supplement: Lvemon verbena extract — Each capsule contained 200 mg of lemon verbena extract 2 capsules/day, 14 days
  Arms: Lemon Verbena extract
Dietary Supplement: maltodextrin — Each capsule contained 0 mg of lemon verbena extract 2 capsules/day, 14 days
  Arms: Placebo

SUMMARY:
In the present study, investigators investigated whether supplementation with lemon verbena extract (LVE) could improve muscle damage and biochemical indicators after exhaustive exercise challenge. Based on maximum jump heights, 60 subjects (30 males and 30 females) were equally divided into a placebo group (0 mg/human/day) and an LVE supplement group (400 mg/human/day), with gender-equal distribution. All subjects started supplementation 10 days before exhaustive exercise and continued it until all tests were completed. Before the intervention, after the exhaustive exercise, and on the following 3 days, the participants underwent 12-minute Cooper running/walking; blood collection; assessments of pain, muscle stiffness, maximum jump heights, and isometric maximum muscle strength; and anaerobic strength tests.

ELIGIBILITY:
Inclusion Criteria:

* health
* Must be able to swallow tablets

Exclusion Criteria:

* non-smokers
* no musculoskeletal
* medical
* metabolic disease
* women not on the reproductive cycle
* high blood pressure, asthma
* skeletal neuromuscular injuries in the upper or lower extremities

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
inflammation of IL-6 level | 10 days
  To assess inflammation indicators, volunteers fasted for at least 8 hours before performing muscle exhaustion exercises. At designated time points in the recovery period, including baseline (0) and 3h, 24h, and 48 after exercise, blood samples were collected with brachial venous catheters. Assess serum IL-6 levels (pg/ml) to monitor physiological fitness. Used commercial kit human IL-6 immunoassay (R&D system, Minnesota, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
Clinical Biochemistry of CK level | 10 days
  To assess muscle damage, volunteers fasted for at least 8 hours before performing muscle exhaustion exercises. At designated time points in the recovery period, including baseline (0) and 3h, 24h, and 48 after exercise, blood samples were collected with brachial venous catheters. Serum CK (U/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Stress hormones 8-Hydroxy-2'-Deoxyguanosine (8-OHdG) in Urine | 10 days
  Subjects' urine was collected 24 hours after the exhaustive exercise for analysis. Used commercial kit human 8-OHdG (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
Assessment of muscle stiffness | 10 days
  3 h, 24h, 48h after exhausting exercise, use Myoton machine to evaluate muscle stiffness (N/m) (Myoton, Tallinn, Estonia)
Visual Analogue Scale (VAS) evaluation | 10 days
  3 h, 24h, 48h after exhausting exercise, use VAS questionnaire to record muscle pain. the minimum is 0 and maximum is 10, and whether higher scores mean more pain

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chang Huang, Ph.D, Principal Investigator — PI
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Lee MC, Hsu YJ, Ho CS, Chang CH, Liu CW, Huang CC, Chiang WD. Evaluation of the Efficacy of Supplementation with Planox(R) Lemon Verbena Extract in Improving Oxidative Stress and Muscle Damage: A Randomized Double-Blind Controlled Trial. Int J Med Sci. 2021 May 3;18(12):2641-2652. doi: 10.7150/ijms.60726. eCollection 2021. PMID 34104096